CLINICAL TRIAL: NCT01951482
Title: Bevacizumab+Pemetrexed/Platinum Versus Pemetrexed/Platinum as First-line Therapy in EGFR/ALK Negative Non-squamous Non-small Cell Lung Cancer Patients With Brain Metastases: a Multicenter, Randomized, Controlled, Phase 3 Study
Brief Title: Pemetrexed/Platinum With or Without Bevacizumab in Brain Metastases From Patients With EGFR/ALK Negative Non-Squamous Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li-kun Chen, medical doctor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC brain metastasis 02
Record Dates: First submitted 2013-09-16; First posted 2013-09-26 (Estimated); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Non Squamous Non-small Cell Lung Cancer; Brain Metastases; Bevacizumab
MeSH Terms: conditions — Brain Neoplasms | interventions — Pemetrexed; Platinum; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bevacizumab plus Pemetrexed/platinum (Experimental): bevacizumab (7.5mg/kg, intravenously on day 1 of each 3-week cycle) plus pemetrexed-platinum chemotherapy (pemetrexed 500mg/m2 combined with cisplatin 75mg/m2 or nedaplatin 80mg/m2 intravenously on day 1 of each 3-week cycle) for four to six cycles, followed by bevacizumab plus pemetrexed maintenance every 3 weeks.
  Interventions: Drug: Bevacizumab and Pemetrexed/platinum
- Pemetrexed/platinum (Active Comparator): pemetrexed 500mg/m2 combined with cisplatin 75mg/m2 or nedaplatin 80mg/m2 intravenously on day 1 of each 3-week cycle for four to six cycles, followed by pemetrexed maintenance every 3 weeks.
  Interventions: Drug: Pemetrexed/Platinum

INTERVENTIONS:
Drug: Pemetrexed/Platinum — pemetrexed 500mg/m2 combined with cisplatin 75mg/m2 or nedaplatin 80mg/m2 intravenously on day 1 of each 3-week cycle for four to six cycles, followed by pemetrexed maintenance every 3 weeks.
  Arms: Pemetrexed/platinum
Drug: Bevacizumab and Pemetrexed/platinum — bevacizumab (7.5mg/kg, intravenously on day 1 of each 3-week cycle) plus pemetrexed-platinum chemotherapy (pemetrexed 500mg/m2 combined with cisplatin 75mg/m2 or nedaplatin 80mg/m2 intravenously on day 1 of each 3-week cycle) for four to six cycles, followed by bevacizumab plus pemetrexed maintenance every 3 weeks.
  Arms: Bevacizumab plus Pemetrexed/platinum

SUMMARY:
This is a multi-center phase 3 randomized controlled study to assess the efficacy of Pemetrexed/platinum with or without Bevacizumab on patients with brain metastasis from non-small cell lung cancer(NSCLC) harboring EGFR/ALK wild type by intracranial PFS(iPFS), also PFS ,ORR, DCR and OS. The safety is evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed non-squamous non-small cell lung cancer (Patients with NSCLC who are newly diagnosed or treated with brain metastases who are asymptomatic or whose intracranial hypertension symptoms are relieved after dehydration treatment, and whose baseline examinations show EGFR wild type (tissue specimen or blood specimen) and ALK negative (tissue specimen);
2. Patients with MRI-confirmed brain metastasis and ≥3 brain lesions; or patients with 1-2 brain lesions but not suitable for local treatment or refusing local treatment. At least one of the brain lesions must be >5 mm in diameter.
3. Age 18-75 years old;
4. Physical condition ECOG score (PS) 0-1;
5. The patient's major organ functions are normal, that is, they meet the following criteria: white blood cells count ≥ 4.0x109/L, neutrophil cells count ≥1.5x109/L, hemoglobin ≥100g/L, serum bilirubin ≤1.5 times the upper limit of normal, transaminase ≤2.5 times the upper limit of normal, if there is liver metastasis, less than 5 times the upper limit of normal; serum creatinine is less than 1.5 times the upper limit of normal, or creatinine clearance is greater than 50ml/min and urine protein is <2+. Patients with baseline urine protein ≥2+ should collect 24-hour urine and prove that the 24-hour urine protein quantitative test is ≤1g.
6. Expected survival time is greater than 12 weeks;
7. Women of childbearing age must undergo a pregnancy test (serum or urine) within 7 days before enrollment, and the result must be negative, and they must be willing to use appropriate contraceptive methods during the trial and within 8 weeks after the last administration of the trial drug. For men, they must agree to use appropriate contraceptive methods during the trial and within 8 weeks after the last administration of the trial drug or have undergone surgical sterilization;
8. Ability to comply with study and follow-up procedures;
9. The patient understands and voluntarily signs the written informed consent.

Exclusion criteria:

Patients who meet any of the following exclusion criteria are not eligible for this trial:

1. Mixed non-small cell and small cell carcinoma, or mixed adenosquamous carcinoma with squamous cells as the main component;
2. Before selection3 A history of hemoptysis within the past month, that is, coughing up at least half a teaspoon of blood;
3. Brain metastases with bleeding;
4. Imaging shows evidence of tumor invasion of large blood vessels. The investigator or radiologist must rule out that the tumor has completely patients with full access, encasement, or invasion into the lumen of large vessels (e.g., pulmonary artery or superior vena cava);
5. Before selection 28 Underwent major surgery (including thoracotomy) within 1 day, suffered major trauma, or patients who are expected to require major surgery during study treatment;
6. First-time bevacizumab/Before placebo treatment48 Minor surgical procedures (including port placement) within 24 hours PICC except);
7. Currently or recently (before receiving first dose of bevacizumab10 Aspirin use (>325 mg/Days) or other nonsteroidal anti-inflammatory drugs known to inhibit platelet function;
8. Currently or recently (before receiving first dose of bevacizumab10 within 2 days) take full dose orally or parenterally anticoagulants or thrombolytics are used for treatment. Prophylactic use of anticoagulants is allowed in patients with deep venous catheters;
9. History or examination findings suggest an inherited bleeding tendency or coagulopathy. Patients with impaired blood flow and thus potentially increased risk of bleeding;
10. Uncontrolled high blood pressure (systolic blood pressure>150 mmHg and/or diastolic blood pressure>100 mmHg);
11. Patients with previous hypertensive crisis or hypertensive encephalopathy;
12. Clinically significant (e.g., active) cardiovascular disease, including but not limited to CVA or TIA (enter before election ≤6 months), myocardial infarction (≤6 months), unstable angina, New York Heart Disease Association Classification ≥II congestive heart failure, requiring medication during the study and may severe arrhythmias that interfere with study treatment or cannot be controlled by medication;
13. Before randomization6 Significant vascular disease within 1 month (including but not limited to active vascular disease requiring surgical repair)aneurysm or recent arterial thrombosis) or thrombotic disease;
14. Non-healing wounds, active peptic ulcers, or fractures;
15. In the selected6 History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 1 month;
16. During the study and after the last dose of bevacizumab within 6 months, with an intact uterus (past twenty four 1 month after menopause), but not using effective contraceptive methods (if combined contraception is not contraindicated Women who used oral contraceptives, intrauterine devices, barrier methods combined with spermicidal gels, or sterilization in the setting of background chemotherapy. Men who do not agree to use effective contraceptive methods;
17. Pregnant and breastfeeding women;
18. Have received any other investigational drug treatment or participated in another clinical trial within 28 days before enrollment;
19. Known hypersensitivity to bevacizumab or any of its excipients and any chemotherapy drug components;
20. Signs of ongoing or active infection requiring intravenous antibiotics, other medical, neurological or metabolic dysfunction, physical examination findings or laboratory test results showing signs of appropriate suspected disease or symptoms that contraindicate the use of the study drug or put the patient at high risk for treatment-related complications;
21. Diagnosed with tracheal-Esophageal fistula;
22. Before randomization5 Years of suffering NSCLC Other malignancies, except for fully treated cervical cancer carcinoma of the uterus, basal cell or squamous cell skin cancer, localized prostate cancer after radical mastectomy, radical mastectomy after ductal carcinoma in situ.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
Compare iPFS(intracranial progression free survival) in two arms | 3 Years

SECONDARY OUTCOMES:
Response rate(CR&PR) | 3 years
safety | 1-year
  adverse events (AEs) were evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events (version 4.0).

OTHER OUTCOMES:
PFS: progress free survival | 3 years
OS: overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: li-kun Chen, Doctor, Study Director — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University of Cancer Center, Guangzhou, Guangdong, China